CLINICAL TRIAL: NCT05092217
Title: Tirelizumab Plus Surgery vs Surgery Alone for Recurrent Nasopharyngeal Carcinoma：a Prospecitve, Parallel, Phase II, Randomized Clinical Trial
Brief Title: Tirelizumab Plus Surgery vs Surgery Alone for Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Dehui Wang, Professor, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rNPC-2021-Dehui Wang
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Recurrent Nasopharyngeal Carcinoma; Tirelizumab; Immunotherapy; Endoscopic surgery; Survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirelizumab plus salvage surgery (Experimental): Tirelizumab: Tirelizumab treatment after salvage surgery. Salvage surgery: endoscopic nasopharyngectomy for recurrent nasopharyngeal carcinoma
  Interventions: Drug: Tirelizumab; Procedure: salvage surgery
- salvage surgery alone (Active Comparator): Salvage surgery: endoscopic nasopharyngectomy for recurrent nasopharyngeal carcinoma
  Interventions: Procedure: salvage surgery

INTERVENTIONS:
Drug: Tirelizumab — Tirelizumab: 200 mg, intravenous injection over 60 minutes (Q3W); Tirelizumab should be applied since 2-6 weeks after surgery until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, investigator decision, or 1 year.
  Other Names: PD-1 antibody
  Arms: Tirelizumab plus salvage surgery
Procedure: salvage surgery — Endoscopic nasopharyngectomy for recurrent nasopharyngeal tumor

SUMMARY:
Through open-label, single-center, randomised clinical trials, we intend to demonstrate that PD-1 treatment added to salvage surgery could further decrease the rate of disease progression and improve the survival outcome of patients with locally recurrent nasopharyngeal carcinoma compared with those treated with salvage surgery alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed recurrent nasopharyngeal carcinoma
2. The recurrence time is more than 6 months from the end of radiotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. According to the TNM staging criteria of nasopharyngeal carcinoma (AJCC, 8th Edition, 2017), rT1, rT2, rT3, and rT4 patients who can be completely resected by surgery as assessed by the surgical team.
5. Resectable recurrent regional lymph node diseases (recurrent N1-3) without prevertebral fascia, cervical vertebrae, or common/internal carotid artery involvement.
6. Given written informed consent.

Exclusion Criteria:

1. Has severe medical disorder, important organ dysfunction, and/or a substantial history of mental illness.
2. Has known subjects with other malignant tumors.
3. Has participated in other drug trials within 3 months of planned start of study treatment.
4. Received a systematic or local glucocorticoid therapy within 4 weeks of planned start of study treatment.
5. Suffered from diseases need long-term treatment with immunosuppressive drugs, or required systematic or local glucocorticoid therapy with immunosuppressive doses.
6. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) agent.
7. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy). Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
8. Has a known history of human immunodeficiency virus (HIV), has hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
9. Has received a live vaccine within 4 weeks of planned start of study treatment.
10. Pregnancy or breast feeding.
11. Cannot complete regular follow-up.
12. Local recurrence of nasopharyngeal carcinoma with distant metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 2 years
  Defined as the time interval from randomization to the observation of disease progression or the occurrence of death from any cause

SECONDARY OUTCOMES:
Overall survival(OS) | 2 years
  Defined as the time interval from randomization to death due to any cause.
Locoregional failure-free survival(LRRFS) | 2 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit
Distant metastasis-free survival(DMFS) | 2 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Incidence of treatment related complications | 2 years
  Incidence of treatment related complications of tirelizumab or surgical treatment during follow-up

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li W, Wang T, Xu H, Liu Q, Zhang H, Yang Y, Sun X, Yu H, Gu Y, Li H, Ding H, Wang D. Tislelizumab as adjuvant therapy following endoscopic surgery for resectable recurrent nasopharyngeal carcinoma: a randomized clinical trial. J Immunother Cancer. 2025 May 24;13(5):e011998. doi: 10.1136/jitc-2025-011998. PMID 40413023